CLINICAL TRIAL: NCT05986526
Title: Pulmonary Vein Isolation With Pulsed-Field Ablation With Versus Without Posterior Wall Ablation in Patients With Symptomatic Persistent Atrial Fibrillation - A Multi-Center Randomized Clinical Trial: The PIFPAF-PFA Study
Brief Title: The PIFPAF-PFA Study
Acronym: PIFPAF-PFA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00885
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Pulmonary vein isolation; Pulsed field ablation; Left atrial posterior wall isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation without posterior wall ablation (Active Comparator): Pulmonary vein isolation without left atrial posterior wall ablation
  Interventions: Procedure: Pulmonary vein isolation without posterior wall ablation
- Pulmonary vein isolation with posterior wall ablation (Active Comparator): Pulmonary vein isolation with left atrial posterior wall ablation
  Interventions: Procedure: Pulmonary vein isolation with posterior wall ablation

INTERVENTIONS:
Procedure: Pulmonary vein isolation without posterior wall ablation — Pulmonary vein isolation with Pulsed field ablation without left atrial posterior wall ablation. At the end of the procedure, an implantable cardiac monitor will be implanted for the purpose of continuous arrhythmia monitoring
  Arms: Pulmonary vein isolation without posterior wall ablation
Procedure: Pulmonary vein isolation with posterior wall ablation — Pulmonary vein isolation with Pulsed field ablation with left atrial posterior wall ablation. At the end of the procedure, an implantable cardiac monitor will be implanted for the purpose of continuous arrhythmia monitoring
  Arms: Pulmonary vein isolation with posterior wall ablation

SUMMARY:
Pulmonary vein isolation (PVI) is very effective for rhythm control in patients with paroxysmal atrial fibrillation (AF), but less successful in patients with persistent AF. Adding posterior wall ablation (PWA) to PVI is among the most promising ablation strategies to improve arrhythmiafree outcome in patients with persistent AF. Patients with left atrial posterior wall scar may benefit most from adding PWA to PVI. With previous ablation technology, posterior wall isolation (PWI) was difficult to achieve and increased the risk of procedural complications. With pulsed-field ablation (PFA), a technology is now available which is both very effective and safe for complete ablation of the posterior wall. The aim of this trial therefore is to compare the efficacy and procedural safety of two ablation strategies for the treatment of persistent AF using PFA: PVI only versus PVI with added PWA. The endpoint of atrial arrhythmia recurrence within 12 months will be assessed by an implantable cardiac monitor (ICM) with remote monitoring capabilities.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent atrial fibrillation documented on a 12 lead ECG, Holter monitor or implantable cardiac device within last 2 years of enrollment
2. Persistent atrial fibrillation is defined as a sustained episode lasting > 7 days
3. Candidate for ablation based on current atrial fibrillation guidelines
4. Continuous anticoagulation with Vitamin-K-Antagonists or a NOAC for ≥4 weeks prior to the ablation; or a transesophageal echocardiography and/or CT scan that excludes left atrial thrombus ≤48 hours before the ablation procedure
5. Age of 18 years or older on the date of informed consent
6. Signed informed consent

Exclusion Criteria:

1. Previous left atrial ablation or left atrial surgery
2. Left atrial diameter >60 mm in the parasternal long axis
3. Patients with paroxysmal atrial fibrillation
4. Patients with persistent atrial fibrillation lasting >3 years
5. AF due to reversible causes (e.g. hyperthyroidism, cardiothoracic surgery)
6. Intracardiac thrombus
7. Pre-existing pulmonary vein stenosis or pulmonary vein stent
8. Pre-existing hemidiaphragmatic paralysis
9. Contraindication to anticoagulation or radiocontrast materials
10. Prior mitral valve surgery
11. Severe mitral regurgitation or moderate/severe mitral stenosis
12. Myocardial infarction during the 3-month period preceding the consent date
13. Ongoing triple antithrombotic/anticoagulation therapy
14. Cardiac surgery during the 3-month interval preceding the informed consent date or scheduled cardiac surgery/ transcatheter aortic valve implantation
15. Significant congenital heart defect (including atrial septal defects or pulmonary vein abnormalities but not including a patent foramen ovale)
16. NYHA class III or IV congestive heart failure
17. Left ventricular ejection fraction (LVEF) <35%
18. Hypertrophic cardiomyopathy (wall thickness >1.5 cm)
19. Significant chronic kidney disease (eGFR <30 ml/min)
20. Uncontrolled hyperthyroidism
21. Cerebral ischemic event (stroke or TIA) during the 6-month interval preceding the informed consent date
22. Ongoing systemic infections
23. History of cryoglobulinemia
24. Cardiac amyloidosis
25. Pregnancy (to exclude pregnancy a blood test (HCG) is performed in women < 50 years before inclusion)
26. Life expectancy less than one year per physician opinion
27. Currently participating in any other clinical trial, which may confound the results of this trial
28. Unwilling or unable to comply fully with the study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2028-02-13 (Estimated)

PRIMARY OUTCOMES:
Time to first recurrence of any atrial tachyarrhythmia | Days 91 to 365 post-ablation
  Time to first recurrence of atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL] or atrial tachycardia [AT]) between days 91 and 365 post ablation as detected on an implantable cardiac monitor (ICM). AF, AFL or AT will qualify as a recurrence after ablation if it lasts 120 seconds or longer on the ICM (the minimum programmable episode interval)

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events: Cardiac tamponade | Days 0 to 90 post-ablation
  Number of patients with cardiac tamponade requiring drainage after PVI
Incidence of treatment-emergent adverse events: Persistent phrenic nerve palsy | Days 0 to 90 post-ablation
  Number of patients with persistent phrenic nerve palsy lasting >24 hours after PVI
Incidence of treatment-emergent adverse events: Serious vascular complication | Days 0 to 90 post-ablation
  Number of patients with serious vascular complications requiring intervention after PVI
Incidence of treatment-emergent adverse events: Stroke or TIA | Days 0 to 90 post-ablation
  Number of patients with stroke or TIA after PVI
Incidence of treatment-emergent adverse events: Atrioesophageal fistula | Days 0 to 90 post-ablation
  Number of patients with atrioesophageal fistula after PVI
Incidence of treatment-emergent adverse events: Death | Days 0 to 90 post-ablation
  Number of patients with fatal outcome/death after PVI
Total procedure time | Day 0, during procedure
  Procedural endpoint
Total left atrial indwelling time | Day 0, during procedure
  Procedural endpoint
Total fluoroscopy time | Day 0, during procedure
  Procedural endpoint
Total radiation dose | Day 0, during procedure
  Procedural endpoint
Change in hs-Troponin on day 1 post-ablation | Day 1 post-ablation
  Procedural endpoint
Pre-ablation 3D electro-anatomical mapping: Number of participants with scar as a region that demonstrated reproducibly an area of > 0.5×0.5 cm on the posterior wall with voltage less than 0.5 mV | Day 0, shortly before ablation
  Procedural endpoint
Post-ablation 3D electro-anatomical mapping: Proportion of isolated veins | Day 0, shortly after ablation
  Procedural endpoint
Post-ablation 3D electro-anatomical mapping: Proportion of isolated carinas | Day 0, shortly after ablation
  Procedural endpoint
Post-ablation 3D electro-anatomical mapping: Lesion size | Day 0, shortly after ablation
  Procedural endpoint
Post-ablation 3D electro-anatomical mapping: Posterior wall ablation success rate | Day 0, shortly after ablation
  Procedural endpoint
Time to first recurrence of any atrial tachyarrhythmia in patients with versus without left atrial posterior wall scar | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Time to first recurrence of any atrial tachyarrhythmia in patients with left atrial posterior wall scar and posterior wall ablation versus without posterior wall ablation | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Percentage of time with cardiac arrhythmia (arrhythmia burden) for each participant between days 0-90 evaluated based on continuous ICM | Day 0 to 90 post-ablation
  Secondary endpoint during follow-up
Percentage of time with cardiac arrhythmia (arrhythmia burden) for each participant between days 91-365 evaluated based on continuous ICM | Day 91 to 365 post-ablation
  Secondary endpoint during follow-up
Percentage of time with cardiac arrhythmia (arrhythmia burden) for each participant between days 365 until explantation or end of life (EOL) of the ICM | Day 365 post-ablation to explantation of ICM or end of life of ICM (up to 4 years after implantation of ICM)
  Secondary endpoint during follow-up
Correlation of AF burden to symptoms and quality of life changes | Day 0 and months 3 and 12 post-ablation
  Secondary endpoint during follow-up; Quality of life wil be measured with the EQ-5D-5L questionnaire where higher scores mean better outcomes; Symptoms will be measured with the AFEQT (Atrial Fibrillation Effect on Quality-of-life) questionnaire where higher scores mean worse outcomes
Reduction of percentage of time with cardiac arrhythmia (AF burden) by > 90% post ablation procedure | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Comparison of the prevalence of the type of arrhythmia recurrence during follow-up being AF or organized atrial arrhythmias (AFL or AT) | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Time to first recurrence of atrial tachyarrhythmia between days 91 and 365 evaluated based on continuous ICM in patients with presence of scar on the PW based on the preablation voltage map versus patients with no scar on the PW | Day 91 to 365 post-ablation
  Secondary endpoint during follow-up
Number of participants with persistent or paroxysmal AF during follow-up | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Average heart rate as recorded by the ICM in months 1, 2 and 3 after ablation | Months 1, 2 and 3 after ablation
  Secondary endpoint during follow-up
Proportion of patients admitted to the hospital or emergency room because of documented recurrence of atrial arrhythmias | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Proportion of patients undergoing a repeat ablation procedure because of documented recurrence of atrial arrhythmias | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Number of participants reinitiating of antiarrhythmic drugs during follow-up | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Number of participants with electrical cardioversion during follow-up | Day 0 to 36 months post-ablation
  Secondary endpoint during follow-up
Number of reconnected pulmonary veins evaluated during redo procedures | During redo procedures between day 1 to 36 months post-ablation
  Secondary endpoint during follow-up
Sites of reconnection (anterior, posterior, superior, inferior) of the pulmonary veins evaluated during redo procedures | During redo procedures between day 1 to 36 months post-ablation
  Secondary endpoint during follow-up
Size of antral scar area (cm²) of the pulmonary veins evaluated during redo procedures | During redo procedures between day 1 to 36 months post-ablation
  Secondary endpoint during follow-up
Number of reconnected posterior walls evaluated during redo procedures | During redo procedures between day 1 to 36 months post-ablation
  Secondary endpoint during follow-up
Sites of reconnection of the posterior wall evaluated during redo procedures | During redo procedures between day 1 to 36 months post-ablation
  Secondary endpoint during follow-up
Size of the scar area (cm²) of the posterior wall evaluated during redo procedures | During redo procedures between day 1 to 36 months post-ablation
  Secondary endpoint during follow-up
Evolution of Quality of Life after 3 and 12 months | Day 0 and months 3 and 12 post-ablation
  Secondary endpoint during follow-up; Quality of life wil be measured with the EQ-5D-5L questionnaire where higher scores mean better outcomes
Number of participants with stroke including TIA after 3, 12, 24 and 36 months | Months 3, 12, 24 and 36 post-ablation
  Secondary endpoint during follow-up
Number of participants with cardiovascular or non-cardiovascular death after 3, 12, 24 and 36 months | Months 3, 12, 24 and 36 post-ablation
  Secondary endpoint during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Roten, MD, Principal Investigator — Inselspital, University Hospital Bern
Locations (6):
- Switzerland (6):
  - Cantonal Hospital Baden, Baden
  - University Hospital Basel, Basel
  - Inselspital, University Hospital Bern, Bern
  - University Hospital Lausanne, Lausanne
  - Cantonal Hospital St. Gallen, Sankt Gallen
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes